CLINICAL TRIAL: NCT06726603
Title: Trends in Pregnancy Outcomes Beyond 20 Weeks Gestational Age in Assisted Reproductive Technology Conceived Pregnancies in BC
Brief Title: Trends in Pregnancy Outcomes Beyond Twenty Weeks Gestational Age in Assisted Reproductive Technology Conceived Pregnancies in British Columbia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mohamed Bedaiwy, Principle Investigator, University of British Columbia
Other Study IDs: H20-00461-A
Record Dates: First submitted 2020-04-29; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2021-02

CONDITIONS: Postpartum Infection
Keywords: Low Birthweight (<2500g); Maternal hospital readmission; Admission to NICU; APGAR Score <6; Cord arterial gas pH<7; premature Birth; Small for gestational Age at Delivery; Perinatal death; Emergency department visit; Gestational Diabetes; Gestational Hypertension; Pre-Eclampsia; HELLP Syndrome; Postpartum infection
MeSH Terms: conditions — Premature Birth; Perinatal Death; Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pre-Eclampsia; HELLP Syndrome | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women in BC conceiving by ART: Women in BC with in-province deliveries following pregnancies conceived by assisted reproductive technology occurring between March 1 2008 and April 31 2018 that resulted in singleton live birth or fetal death at >20 weeks.
  Interventions: Procedure: Assisted Reproductive Technology
- Women in BC conceiving spontaneously: Women in BC with in-province deliveries following pregnancies conceived spontaneously occurring between March 1 2008 and April 31 2018 that resulted in singleton live birth or fetal death at >20 weeks.

INTERVENTIONS:
Procedure: Assisted Reproductive Technology — Assisted Reproductive Technology for the purposes of this study include IVF and IVF+ICSI. Ovulation induction methods are not considered Assisted Reproductive Technology
  Groups: Women in BC conceiving by ART

SUMMARY:
Examining outcomes beyond 20 weeks gestational age in pregnancies conceived by ART compared to spontaneously conceived pregnancies

1. To determine if a difference in outcomes for pregnancies beyond 20 weeks gestational age exists between ART-treated and spontaneous conception populations in BC. Specifically, the investigators will examine the prevalence for gestational diabetes, gestational hypertension, premature deliveries, low birth weight, miscarriages, maternal length of stay in hospital, NICU admissions, APGAR scores<6, and arterial cord gas pH<7.
2. To examine the trend of outcomes beyond 20 weeks GA associated with ART by calendar year from March 2008 to April 2018.

The research literature from other study populations suggest the prevalence of pregnancy complications are higher amongst women with ART-treated deliveries. Specifically, there is a trend towards higher rates of gestational diabetes, pregnancy induced hypertension, premature deliveries, low birthweight deliveries, perinatal deaths and maternal length of stay in hospital after delivery. The challenge lies in determining the degree of difference and the trend.

Given the relatively older age of conception in BC, the investigators hypothesize that the aforementioned complications may in fact be higher in both the spontaneous conception and ART-treated groups. That being said, the investigators suspect the ART group is likely to still have a higher rates of gestational diabetes, hypertension, premature deliveries, low birthweight, and miscarriages.

DETAILED DESCRIPTION:
The investigators intend to conduct a retrospective cohort study examining differences in pregnancy outcomes after 20 weeks GA in ART-treated versus fertile women.

The study population will consist of women in BC with in-province deliveries occurring between March 1 2008 and April 31 2018 that resulted in singleton live birth or fetal death at >20 weeks. Only fertile women conceiving their index pregnancy by assisted reproductive technology (ART) will be included. Multiparous women and women with multiple gestation deliveries will be excluded. Also, any women missing data including gravida, parity, age, date of birth, neonatal birth weight, neonatal APGARs, neonatal live birth versus stillbirth Data will be collected from the perinatal services BC database, following approval. A biostatistician will be employed to help utilize the data requested.

Obstetric and Fetal outcome measures of prematurity (<37 weeks GA), low birthweight (<2500g), small for gestational age (in live births), perinatal death (fetal death >20 weeks to death of newborn up to 7 days post-delivery), prolonged maternal length of stay in hospital following delivery (>3 days), and maternal hospital readmission (rehospitalization 0-60 days after delivery plus emergency department of observation stay visits 0-7 days after delivery), gestational diabetes (insulin and non-insulin dependent), gestational hypertension (>140/90 after 20 weeks GA), pre-eclampsia HELLP Syndrome, Postpartum infection, admission to NICU, APGAR score <6, cord arterial gas pH <7. Chi square statistics will be used to evaluate statistical differences in binary outcomes among fertile and ART-treated groups while ANOVA tests will be implemented to evaluate differences in continuous outcomes. Multivariable models will be adjusted for potential confounders including maternal age (30, 31-34, 35-37, 38-40, >40), smoking (yes/no), chronic hypertension (yes/no), pre-pregnancy diabetes (type 1 and type 2), pre-pregnancy BMI equal to or greater than 30.

ELIGIBILITY:
Inclusion Criteria:

* Women in BC with in-province deliveries occurring between March 1 2008 and April 31 2018 that resulted in singleton live birth or fetal death at >20 weeks
* Only fertile and women conceiving their index pregnancy by assisted reproductive technology (ART) will be included.

Exclusion Criteria:

* Multiparous women and women with multiple gestation deliveries will be excluded
* any women missing data including gravida, parity, age, date of birth, neonatal birth weight, neonatal APGARs, neonatal live birth versus stillbirth will be excluded

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women in BC with in-province deliveries (following naturally conceived or assisted reproductive technologies) occurring between March 1 2008 and April 31 2018 that resulted in singleton live birth or fetal death at >20 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Pregnancy complications beyond 20 weeks gestation age | From point at which patient is 20 weeks gestational age to one month postpartum
Pre-eclampsia | From point at which patient is 20 weeks gestational age to one month postpartum
  Blood pressure of 140/90 mmHg or higher and symptoms or signs of ongoing damage to internal organs
Gestational hypertension | From point at which patient is 20 weeks gestational age to one month postpartum
  Blood pressure of 140/90 mmHg or higher and no symptoms or signs of ongoing damage to internal organs
HELPP syndrome | From point at which patient is 20 weeks gestational age to one month postpartum
  Evidence of hemolysis, elevated liver enzymes, Low platelets
Low birth weight of infant | From point at which patient is 20 weeks gestational age to one month postpartum
  <2500 grams
small for gestational age | From point at which patient is 20 weeks gestational age to one month postpartum
  A weight below the 10th percentile for the gestational age.
Gestational diabetes | This outcome is measured from point at which patient is 20 weeks gestational age to one month postpartum
Low APGAR score | From point at which patient is 20 weeks gestational age to one month postpartum, depends on delivery timing
  AGPAR score less than 6 at time of live birth delivery
Cord arterial pH< 7 | From point at which patient is 20 weeks gestational age to one month postpartum
  At time of delivery of neonate
NICU admission | From point at which patient is 20 weeks gestational age to one month postpartum
  Admission to NICU
perinatal death | From point at which patient is 20 weeks gestational age to 7 days post-delivery
  fetal death >20 weeks to death of newborn up to 7 days post-delivery

SECONDARY OUTCOMES:
Maternal re-admission to hospital | From delivery to 60 days after maternal delivery
  rehospitalization 0-60 days after delivery plus emergency department of observation stay visits 0-7 days after delivery
Maternal postpartum infection | from delivery to one month postpartum
  infection from pregnancy and/or delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bedaiwy, MD, PhD, Principal Investigator — University of British Columbia